CLINICAL TRIAL: NCT03665376
Title: Feasibility and Efficacy of Enhanced Recovery After Surgery (ERAS) on Length of Stay Among Laparotomy Patients at Mbarara Regional Referral Hospital, Uganda
Brief Title: Feasibility and Efficacy of Enhanced Recovery After Surgery (ERAS) on Length of Stay Among Laparotomy Patients at Mbarara Regional Referral Hospital
Acronym: ERAS-Lap
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mbarara University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MUST16/2017
Record Dates: First submitted 2018-09-05; First posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Laparotomy
MeSH Terms: interventions — Enhanced Recovery After Surgery

STUDY DESIGN:
Intervention Model Description: Participants were randomly allocated into two arms: intervention arm (ERAS) and control arm
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS arm (Experimental): Preoperative: Counseling and education about the ERAS program; Oral intake until 6 hours before the surgery; Carbohydrate drinks load; No mechanical bowel preparation; Antithrombotic prophylaxis (Tinzaparin 3500 IU) Intraoperative: Spinal anaesthesia (15 mg hyperbaric Bupivacaine + 200mcg intrathecal Morphine); Intravenous Ceftriaxone 2g, Metronidazole 500mg / Gentamycin 160mg, Ondansetron 8mg and Dexamethasone 8mg; Crystalloid fluid 10 to 20ml/Kg; Adrenaline 200mcg in each 500 ml of intravenous fluid; Avoidance of abdominal drains; Postoperative: Early oral intake; Nasogastric tube and urinary catheter removed immediately after the surgery; Early enteral nutrition; Chewing gum for 2 to 4 hours after surgery; Oral sips 8 hours postoperatively; Intravenous fluids discontinued at four hours after transfer to the ward.
  Interventions: Dietary Supplement: Carbohydrate drink load; Combination Product: Enhanced Recovery After Surgery (ERAS)
- Control arm (No Intervention): Preoperative: No carbohydrate drink loads, no antithrombotic prophylaxis; Mechanical bowel preparation as needed; Spinal anaesthesia, fluid therapy and antibiotherapy done according to standard hospital practice. The urinary catheter and drains were removed at the discretion of the surgeon. Postoperative: Enteral feeding delayed by the auscultation of bowel sounds. The standard hospital practices involve keeping active the nasogastric tube, fasting patients postoperative, strict bed rest… Pain control was managed with medication of choice by surgeon and anesthesiologist.

INTERVENTIONS:
Dietary Supplement: Carbohydrate drink load — Administration of 5% Dextrose orally as a carbohydrate drink load two hours before surgery and as an oral sips eight hours after the surgery.
  Other Names: 5% Dextrose orally
  Arms: ERAS arm
Combination Product: Enhanced Recovery After Surgery (ERAS) — The ERAS intervention consisted of exposing patients to ERAS protocol of care as described by the ERAS Society® for the entire perioperative period. However, some of these ERAS protocols were modified to our local resources and requirements.
  Other Names: Fast Track Surgery; Multimodal Rehabilitation
  Arms: ERAS arm

SUMMARY:
The main goal of ERAS is to enhance the recovery of patients, and this has secondary effects, such reduced length of hospital stay, minimal postoperative complications and lessen readmission rates. ERAS protocols have been shown to be feasible and safe across the world. Although it has been shown to be effective in the developed settings and can potentially reduce the length of hospital stay, and the cost of healthcare in the perioperative period. The multimodal program of ERAS has been less implemented in the low and middle income African countries. Studies done outside Uganda (Egypt and South Africa) have demonstrated that ERAS program can be feasible and yields favorable outcomes in patients.

DETAILED DESCRIPTION:
The efficacy of ERAS has been demonstrated in resource rich settings but limited evidence is available from resource poor settings. The aim of this study was to determine the feasibility and test efficacy of ERAS in reducing length of post-operative hospital stay and the incidence of postoperative complications compared to the standard of care as the control group.

33 participants above 18 years of age, undergoing laparotomy, were randomly assigned to an intervention (ERAS) arm or to a control (standard surgical care) arm at Mbarara Regional Referral Hospital in Uganda. The ERAS and the control arm had 16 and 17 patients respectively, followed-up 14 days after surgery.

Patients in the ERAS arm had 2.4 days (SD 0.7) of post-operative hospital stay shorter than those in the control arm, p=0.0025 (4.1±0.2 vs 6.5±0.6 respectively). 18.8% of patients in the control arm developed post-operative complications compared to 5.9% in the ERAS arm (Statistical insignificance, p=0.34). ERAS patients passed flatus eight hours earlier than patients in the control arm, and mobilisation out of bed happened 12 hours earlier in the ERAS group p value=0.4.

ERAS is feasible at Mbarara Regional Referral Hospital, and it leads to reduced hospital stay duration but not post-operative complications in laparotomy cases.

ELIGIBILITY:
Inclusion Criteria:

* We enrolled adult patients, 18 years of age and above, scheduled for non-emergency laparotomy.

Exclusion Criteria:

* Patients with age less than 18 years
* Pregnant patients
* Emergency Laparotomy
* American Society of Anesthesiologists (ASA) physical status score greater than 3
* Surgeries other than elective gastrointestinal laparotomy
* Diabetes patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2017-07-30 (Actual); Study Completion 2017-08-15 (Actual)

PRIMARY OUTCOMES:
Length of hospital stay | From the day of surgical operation up to time 14 days
  It is the duration of a single episode of hospitalization measured as time .

SECONDARY OUTCOMES:
Perioperative morbidity and mortality | From the start of surgical intervention to 14 days after discharge from the hospital
  Adverse events or death occurring during or 14 days after the surgical operation
Readmission rate | Within 14 days from the day of discharge from the hospital
  Admission of a patient in the hospital within 14 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Serge M Tshijuke, MD, MMed, Principal Investigator — Kabale University
Locations (1):
- Mbarara Regional Referral Hospital, Mbarara, Uganda